CLINICAL TRIAL: NCT04401397
Title: The Effect of Inpatient Intensive Early Mobilisation Intervention on Length of Hospital Stay, Medical and Functional Recovery and Readmission Rate of Patients After CABG or AVR/MVR: A Randomized Single Blind Controlled Clinical Trial.
Brief Title: Effect of Early Mobilization on Length of Stay, Recovery and Readmission Rate of Patients After CABG or AVR/MVR Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dimitris Chatzitheodorou (Other)
Collaborators: University of Macedonia, Thessaloniki, Greece (Other)
Responsible Party: Sponsor-Investigator, Dimitris Chatzitheodorou, Principal Investigator, Senior Physical Therapist, Papageorgiou General Hospital
Organization: Papageorgiou General Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: PapageorgiouGH
Record Dates: First submitted 2020-05-15; First posted 2020-05-26 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease; Aortic Valve Disease; Mitral Valve Disease
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Disease

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled double-blind 2-group experimental design.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and outcomes assessor will be blinded to the protocol each patient will be treated with. Both intervention and standard care protocols will be implemented by a third party.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early mobilization group (Experimental): Immediately after ICU extubation, enrolled patients will receive an intensive 30-45 minutes, implemented twice a day early mobilization protocol containing psychological empowerment, detailed informative education of patients and close relatives, close monitoring of the recovery course, frequent parameter protocol configuration, high intensity active progressive pulmonary and musculoskeletal exercises and mobility techniques, close monitoring for early identification and measures for prevention and treatment of complications.
  Interventions: Procedure: Intensive early mobilization techniques
- Standard care group (Active Comparator): Enrolled patients will receive the standard hospital mobilization protocol after their admission to the ward, containing standardized basic pulmonary and mobilization techniques of 15 minutes, once a day.
  Interventions: Procedure: Intensive early mobilization techniques

INTERVENTIONS:
Procedure: Intensive early mobilization techniques — Pulmonary techniques: lung mechanics and breathing pattern restoration, mucus clearance techniques, breathing control and cough techniques.
  Musculoskeletal techniques: strengthening and functional exercises, active assistive moving techniques.

SUMMARY:
The present study will investigate the volume and extent of the expected physiological effects of "early mobilization" on the prevention of the clinical illness' detrimental sequelae and on the functional recovery promotion of CABG, AVR and MVR patients. Consequently, it will investigate if the improved health outcomes may limit the number and intensity of complications and thus if it may speed up hospital discharge.

DETAILED DESCRIPTION:
Although the effects of "early mobilization" have been studied mainly in the intensive care unit setting, the findings could be applied to the surgical units' patients too, since they share common physiological and clinical characteristics. In the literature the effectiveness of "early mobilization" in the length of hospital stay and recovery of the patients operated for coronary artery bypass graft and heart valve replacement in the cardiac surgery setting, is unknown.

The term "early mobilization" is not restricted to a time factor procedure but contains the provision of a customized dynamic set of physical therapy techniques which in studies are variably determined in terms of duration, intensity, frequency and content.

The aim of the study is to determine the clinical effectiveness of the intensive early mobilization physical therapy intervention compared with standard care of physical therapy in the cardio-thoracic surgery clinic of Papageorgiou General Hospital of Thessaloniki.

The present study will investigate the volume and extend of the expected physiological effects of "early mobilization" on the prevention of the clinical illness' detrimental sequelae and on the functional recovery promotion, hospital mortality and readmission rate of CABG, AVR and MVR patients. Consequently, it will investigate if the improved health outcomes may limit the number and intensity of complications and thus may speed up hospital discharge. In the first group of the experimental design, patients will be treated with an intensive early mobilization protocol and the patients of the second group will receive a standard care physical therapy treatment. Controlling for the detailed baseline characteristics that will be assessed during medical history at admission, potential bias will be limited from unmeasured confounders of the study.

ELIGIBILITY:
Inclusion Criteria:

* Elective CABG or AVR or MVR surgery
* No previous CABG or valve surgery
* Isolated / multivessel CABG

Exclusion Criteria:

* Current neurological disorders
* Previous cerebral vascular accident with residual neurological deficit significant enough to limit exercise
* Significant limiting comorbidities that would prevent full participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Length of postoperative hospital stay | Up to 6 weeks
  The number of postoperative days that the patients stay in the ward after their surgery procedure and ICU discharge.
Readmission rate | Up to 6 weeks
  The number of discharged patients that will be readmitted in the hospital for a condition of their underlying disease in a 30 days period after surgery.
Number of complications | Up to 6 weeks
  The total number of medical events the patients will develop during their postoperative stay in the ward.
Severity of complications | Up to 6 weeks
  Classification of the complications as "minor" or "major" according to the physicians' expert opinion based on published clinical standards.
Time to regain hemodynamic stability | Up to 6 weeks
  The time in days that is required for the patients to be without inotrope or vasodilator drugs and remain normal and stable in arterial blood pressure, heart rate and blood gas rates.
Two-minute walk test | Up to 6 weeks
  The distance in meters that a patient can walk under the specific test conditions, at the day of discharge.
Functional recovery | Up to 6 weeks
  The time in days that is required for the patients to be autonomous in accessing and using the toilet in their ward.
High cost medical procedures | Up to 6 weeks
  The number of high cost medical procedures the patients will undergo during their postoperative stay in the ward.

SECONDARY OUTCOMES:
Hospital mortality | Up to 6 weeks
  The number of postsurgical hospital deaths.

CONTACTS AND LOCATIONS:
Locations (1):
- Papageorgiou General Hospital, Thessaloniki, Pavlou Mela Municipality, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiarici A, Andrenelli E, Serpilli O, Andreolini M, Tedesco S, Pomponio G, Gallo MM, Martini C, Papa R, Coccia M, Ceravolo MG. An Early Tailored Approach Is the Key to Effective Rehabilitation in the Intensive Care Unit. Arch Phys Med Rehabil. 2019 Aug;100(8):1506-1514. doi: 10.1016/j.apmr.2019.01.015. Epub 2019 Feb 21. PMID 30796918
- [Background] Corcoran JR, Herbsman JM, Bushnik T, Van Lew S, Stolfi A, Parkin K, McKenzie A, Hall GW, Joseph W, Whiteson J, Flanagan SR. Early Rehabilitation in the Medical and Surgical Intensive Care Units for Patients With and Without Mechanical Ventilation: An Interprofessional Performance Improvement Project. PM R. 2017 Feb;9(2):113-119. doi: 10.1016/j.pmrj.2016.06.015. Epub 2016 Jun 23. PMID 27346093
- [Background] Lord RK, Mayhew CR, Korupolu R, Mantheiy EC, Friedman MA, Palmer JB, Needham DM. ICU early physical rehabilitation programs: financial modeling of cost savings. Crit Care Med. 2013 Mar;41(3):717-24. doi: 10.1097/CCM.0b013e3182711de2. PMID 23318489
- [Background] Tsuboi N, Hiratsuka M, Kaneko S, Nishimura N, Nakagawa S, Kasahara M, Kamikubo T. Benefits of Early Mobilization After Pediatric Liver Transplantation. Pediatr Crit Care Med. 2019 Feb;20(2):e91-e97. doi: 10.1097/PCC.0000000000001815. PMID 30489487
- [Background] van Willigen Z, Collings N, Richardson D, Cusack R. Quality improvement: The delivery of true early mobilisation in an intensive care unit. BMJ Qual Improv Rep. 2016 Dec 30;5(1):u211734.w4726. doi: 10.1136/bmjquality.u211734.w4726. eCollection 2016. PMID 28090326
- [Background] Brummel NE, Girard TD, Ely EW, Pandharipande PP, Morandi A, Hughes CG, Graves AJ, Shintani A, Murphy E, Work B, Pun BT, Boehm L, Gill TM, Dittus RS, Jackson JC. Feasibility and safety of early combined cognitive and physical therapy for critically ill medical and surgical patients: the Activity and Cognitive Therapy in ICU (ACT-ICU) trial. Intensive Care Med. 2014 Mar;40(3):370-9. doi: 10.1007/s00134-013-3136-0. Epub 2013 Nov 21. PMID 24257969
- [Background] Li Z, Peng X, Zhu B, Zhang Y, Xi X. Active mobilization for mechanically ventilated patients: a systematic review. Arch Phys Med Rehabil. 2013 Mar;94(3):551-61. doi: 10.1016/j.apmr.2012.10.023. Epub 2012 Nov 2. PMID 23127305
- [Background] Parker A, Sricharoenchai T, Needham DM. Early Rehabilitation in the Intensive Care Unit: Preventing Physical and Mental Health Impairments. Curr Phys Med Rehabil Rep. 2013 Dec;1(4):307-314. doi: 10.1007/s40141-013-0027-9. PMID 24436844
- [Background] Adler J, Malone D. Early mobilization in the intensive care unit: a systematic review. Cardiopulm Phys Ther J. 2012 Mar;23(1):5-13. PMID 22807649
- [Background] Mendez-Tellez PA, Nusr R, Feldman D, Needham DM. Early Physical Rehabilitation in the ICU: A Review for the Neurohospitalist. Neurohospitalist. 2012 Jul;2(3):96-105. doi: 10.1177/1941874412447631. PMID 23983871
- [Background] Morris PE, Griffin L, Berry M, Thompson C, Hite RD, Winkelman C, Hopkins RO, Ross A, Dixon L, Leach S, Haponik E. Receiving early mobility during an intensive care unit admission is a predictor of improved outcomes in acute respiratory failure. Am J Med Sci. 2011 May;341(5):373-7. doi: 10.1097/MAJ.0b013e31820ab4f6. PMID 21358312
- [Background] Needham DM, Korupolu R, Zanni JM, Pradhan P, Colantuoni E, Palmer JB, Brower RG, Fan E. Early physical medicine and rehabilitation for patients with acute respiratory failure: a quality improvement project. Arch Phys Med Rehabil. 2010 Apr;91(4):536-42. doi: 10.1016/j.apmr.2010.01.002. PMID 20382284
- [Background] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Background] Morris PE, Goad A, Thompson C, Taylor K, Harry B, Passmore L, Ross A, Anderson L, Baker S, Sanchez M, Penley L, Howard A, Dixon L, Leach S, Small R, Hite RD, Haponik E. Early intensive care unit mobility therapy in the treatment of acute respiratory failure. Crit Care Med. 2008 Aug;36(8):2238-43. doi: 10.1097/CCM.0b013e318180b90e. PMID 18596631
- [Background] Hopkins RO, Spuhler VJ, Thomsen GE. Transforming ICU culture to facilitate early mobility. Crit Care Clin. 2007 Jan;23(1):81-96. doi: 10.1016/j.ccc.2006.11.004. PMID 17307118
- [Background] Bailey P, Thomsen GE, Spuhler VJ, Blair R, Jewkes J, Bezdjian L, Veale K, Rodriquez L, Hopkins RO. Early activity is feasible and safe in respiratory failure patients. Crit Care Med. 2007 Jan;35(1):139-45. doi: 10.1097/01.CCM.0000251130.69568.87. PMID 17133183
- [Background] Gosselink R, Bott J, Johnson M, Dean E, Nava S, Norrenberg M, Schonhofer B, Stiller K, van de Leur H, Vincent JL. Physiotherapy for adult patients with critical illness: recommendations of the European Respiratory Society and European Society of Intensive Care Medicine Task Force on Physiotherapy for Critically Ill Patients. Intensive Care Med. 2008 Jul;34(7):1188-99. doi: 10.1007/s00134-008-1026-7. Epub 2008 Feb 19. PMID 18283429